CLINICAL TRIAL: NCT04519528
Title: Acute Neurological Complications and Neurodevelopmental Outcome in Children Undergoing Extracorporeal Membrane Oxygenation.
Acronym: NeurECMO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200675; 2020-A01185-34 (Other: IDRCB number)
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Extra Corporeal Membrane Oxygenation
Keywords: Extra corporeal membrane oxygenation; Pediatric patients; Neurological complications; Neurological outcome; Quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Minors who required veno-venous or veno-arterial ECMO, in pediatric intensive care unit at Necker Enfants Malades hospital between 2014 and 2019.
  Interventions: Other: DENVER scale (under 2 years old) or Pediatric Cerebral Performance Category (PCPC) score (over 2 years old); Other: Pediatric Quality of Life Inventory™ (PedsQL)

INTERVENTIONS:
Other: DENVER scale (under 2 years old) or Pediatric Cerebral Performance Category (PCPC) score (over 2 years old) — The DENVER II is a measure of developmental problems in young children. It was designed to assess child performance on various age-appropriate tasks and compares a given child's performance to the performance of other children the same age. The instrument consists of 125 tasks, which broadly reflect the following areas: personal-social, fine motor-adaptive, language, and gross motor.
  The target population corresponds to infants and pre-school age children.
  The POPC and PCPC are global scales based on observer impressions. Scores include 1 for good, 2 for mild disability, 3 for moderate disability, 4 for severe disability, and 5 for vegetative state or coma (6 indicates death).
  Other Names: Neurological assessment
Other: Pediatric Quality of Life Inventory™ (PedsQL) — The PedsQL questionnaire is a modular approach to measuring health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. The PedsQL Measurement Model integrates seamlessly both generic core scales and disease-specific modules into one measurement system. Twenty-three items divided into different functional areas are evaluated: physical (8 items), emotional (5 items), social (5 items) and school (5 items over 4 years old; 3 items before 4 y.o).
  Child self-report and parent proxy report formats of the questionnaire allows self-assessment of child over 5 years old and parents' evaluations. Items can be reverse and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0) with higher scores indicating better quality of life.
  Other Names: Quality of life assessment

SUMMARY:
The purpose of this retrospective study is to describe the different types of acute neurologic complications in children who underwent extracorporeal membrane oxygenation (ECMO), and their risk factors. The research will also assess the child health at 1 year after withdrawal from ECMO and in 2020 in terms of neurological state and quality of life.

DETAILED DESCRIPTION:
Neurological complications are relatively common (around 30%) in patients undergoing extra corporeal membrane oxygenation (ECMO). They can be hemorrhagic or ischemic and are partly due to the difficulty of balancing heparin therapy. Few pediatric studies have estimated the incidence and risk factors for these lesions. In addition, the developmental monitoring and quality of life of these children is not systematic or standardized, and their long-term outcome deserves to be better evaluated.

The purpose of this retrospective study is to describe the different types of acute neurologic complications in children who underwent veno-veinous or veno-arterial ECMO and their risk factors. The study is being conducted at Necker Enfants Malades hospital between 2014 and 2019. The research will also assess the child health at 1 year after withdrawal from ECMO and in 2020 in terms of neurological state and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Children from 0 to 18 years hospitalized in PICU (pediatric intensive care unit) and who underwent veno-venous or veno-arterial extra corporeal membrane oxygenation (ECMO) between 2014 and 2019.
* Adult patients not oppose to participation in research or holders of parental authority of minor patients not opposed to participation in the study.

Exclusion Criteria:

- Other type of assistance than an ECMO (Berlin heart).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Minors from 0 to 18 years hospitalized in pediatric resuscitation of Necker hospital and placed on veno-venous or veno-arterial extra corporeal membrane oxygenation (ECMO) between 2014 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Risk factors of neurological complications | 9 days
  Identification of risk factors of neurological complications acquired under ECMO by significant association between neurological lesions diagnosed on imaging and the co-variables.

SECONDARY OUTCOMES:
Diagnosis of neurological lesions | 9 days
  Description of different types of neurological complications acquired under ECMO with brain CT scan or MRI.
Death | 6 years
  Number of death.
Delay between ECMO withdrawal and death | 6 years
  Children who died after ECMO withdrawal.
Neurological assessment | At one year after ECMO withdrawal, and in 2020
  Score at DENVER scale or Pediatric Cerebral Performance Category (PCPC) score.
Quality of life assessment | At one year after ECMO withdrawal, and in 2020
  Score at Pediatric Quality of Life Inventory™ (PedsQL).

CONTACTS AND LOCATIONS:
Overall Officials: Judith Chareyre, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michel A, Vedrenne-Cloquet M, Kossorotoff M, Thy M, Levy R, Pouletty M, De Marcellus C, Grimaud M, Moulin F, Hully M, Simonnet H, Desguerre I, Renolleau S, Oualha M, Chareyre J. Neurologic Outcomes and Quality of Life in Children After Extracorporeal Membrane Oxygenation. Pediatr Crit Care Med. 2024 Mar 1;25(3):e158-e167. doi: 10.1097/PCC.0000000000003419. Epub 2023 Dec 13. PMID 38088764